CLINICAL TRIAL: NCT07382557
Title: Adaptation and Pilot Testing of a Lung Cancer Screening Decision Aid for Patients From a Safety-Net Healthcare System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-0383
Record Dates: First submitted 2025-06-30; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Needs Assessment: Provider Survey (Aim 1) (Other): Up to 200 physicians and other health professionals
  Interventions: Other: Surveys
- Needs Assessment: Patient/Family member Focus Groups (Aim 1) (Other): Up to 20 participants who speak English or Spanish
  Interventions: Other: Focus groups
- Decision Aid Adaptation (Patient Cognitive Interviews (Aim 1) (Other): Up to 40 participants who speak English or Spanish
  Interventions: Other: Cognitive Interviews
- Pilot Study: Intervention Patients (Aim 2) (Experimental): Up to 50 participants (25 English speakers, 25 Spanish speakers)
  Interventions: Behavioral: Lung cancer screening decision aid video
- Pilot Study: Control Patients (Aim 2) (Placebo Comparator): Up to 50 participants (25 English speakers, 25 Spanish speakers)
  Interventions: Behavioral: Colon cancer screening video

INTERVENTIONS:
Other: Surveys — Investigators will answer surveys about their lung cancer screening practices
  Arms: Needs Assessment: Provider Survey (Aim 1)
Other: Focus groups — Participants will participate in focus groups about information they need in order to decide about lung cancer screening
  Arms: Needs Assessment: Patient/Family member Focus Groups (Aim 1)
Other: Cognitive Interviews — Participants will participate in interviews about their understanding of the adapted video script
  Arms: Decision Aid Adaptation (Patient Cognitive Interviews (Aim 1)
Behavioral: Lung cancer screening decision aid video — Participants take surveys before and after watching the intervention video
  Arms: Pilot Study: Intervention Patients (Aim 2)
Behavioral: Colon cancer screening video — Participants take surveys before and after watching the control video
  Arms: Pilot Study: Control Patients (Aim 2)

SUMMARY:
The goal of the study is to adapt and test a participant decision aid about lung cancer screening for use with patients in theHarris Health System (HHS).

DETAILED DESCRIPTION:
The study has two phases. In the first phase, the investigators will conduct a cultural and linguistic adaptation of a patient decision aid video on lung cancer screening for use with patients with low health literacy in English and Spanish. They will produce adapted decision aid videos and written educational materials about lung cancer screening. They will survey providers about their lung cancer screening practices, conduct focus groups to learn what patients want to know about screening, and perform cognitive interviews with patients to make sure the adapted videos and educational materials are easy to understand.

In the second phase, the investigators will test the adapted lung cancer screening decision aid videos in English and Spanish to determine acceptability and impact of the aids on decision making outcomes. Patients will be randomized to evaluate an adapted video decision aid intervention or a control condition.

ELIGIBILITY:
Inclusion Criteria:

1. 50-80 years of age
2. Current smokers or smokers who have quit less than 15 years ago
3. Speak either English or Spanish
4. No history of lung cancer
5. Family member of someone with a history of smoking AND lung cancer

Exclusion Criteria:

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs). | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vok, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org